CLINICAL TRIAL: NCT06225284
Title: A Randomized Phase II Study of Neoadjuvant Chemotherapy With or Without GnRH Agonist for Premenopausal Triple-negative Early Breast Cancer Patients: ESCALATE Study
Brief Title: Neoadjuvant Chemotherapy With or Without GnRH Agonist for Premenopausal Triple-negative Early Breast Cancer Patients
Acronym: ESCALATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Health and Welfare (Ambiguous); Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202309050MIPB
Record Dates: First submitted 2023-12-10; First posted 2024-01-25 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Triple Negative Breast Cancer; Premenopausal Breast Cancer
Keywords: Neoadjuvant chemotherapy; Triple negative breast cancer; Gonadotropin Releasing Hormone Agonist; Premenopausal Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): After randomization, patients in the experimental arm (Arm A) will receive GnRH agonist injection within 7 days of randomization and during neoadjuvant chemotherapy treatment. The protocol-defined chemotherapy will be given 7 to 14 days after GnRH agonist injection. The choice of GnRH agonist, including goserelin, leuprorelin and triptorelin giving in monthly, three-monthly or sixth-monthly, will be made by per investigator's discretion.
  * Anthracycline-cyclophosphamide combination or Anthracycline-cyclophosphamide combination, dose-dense schedule
  * Taxane (docetaxel or paclitaxel) ± optional platinum (Use of platinum or not will be stratified.)
  * Optional pembrolizumab(Use of pembrolizumab or not will be stratified.)
  Interventions: Drug: Goserelin Acetate 3.6mg、Goserelin Acetate 10.8mg、Leuprolide Acetate 3.75mg、Leuprorelin Acetate 22.5mg、Triptorelin pamoate 11.25mg、Triptorelin pamoate 22.5mg
- Arm B (No Intervention): * Anthracycline-cyclophosphamide combination or Anthracycline-cyclophosphamide combination, dose-dense schedule
  * Taxane (docetaxel or paclitaxel) ± optional platinum (Use of platinum or not will be stratified.)
  * Optional pembrolizumab(Use of pembrolizumab or not will be stratified.)

INTERVENTIONS:
Drug: Goserelin Acetate 3.6mg、Goserelin Acetate 10.8mg、Leuprolide Acetate 3.75mg、Leuprorelin Acetate 22.5mg、Triptorelin pamoate 11.25mg、Triptorelin pamoate 22.5mg — After randomization, patients in the experimental arm (Arm A) will receive GnRH agonist injection within 7 days of randomization and during neoadjuvant chemotherapy treatment. The choice of GnRH agonist, including goserelin, leuprorelin and triptorelin giving in monthly, three-monthly or sixth-monthly, will be made by per investigator's discretion.
  Arms: Arm A

SUMMARY:
Breast cancer (BC), especially premenopausal, is emerging rapidly in East Asia in recent 20 years. Half of the breast cancer patients in Asia are younger than 50 years of age. In general, younger or premenopausal patients are associated with poorer prognosis.

Premenopausal patients have higher estrogen levels than those in older (postmenopausal) patients. Estrogen is known to suppress anti-tumor T cell response and leading to tumor progression in different animal models (Clin Cancer Res 2016 22:6204), including lung cancer, melanoma, ovarian cancer. One of the mechanisms that contributes to estrogen's suppression of T cell function is via the mobilization of myeloid-derived suppressor cells (MDSC). Targeting ER signaling with hormonal therapy can abolish MDSC mobilization, and sensitize tumor cells to antigen specific T cell or NK cell killing (Cancer Discovery 2018 7:72 2017). These study results further support the hypothesis that, E2 is associated with immunosuppressive effect, and may contribute to the suppression of immune surveillance in young female breast cancer patients. These results suggest that E2 may suppress anti-tumor immunity, and E2 reduction improve the anti-tumor immunity. In our preliminary works, the investigators found higher dose (equivalent to premenopausal women serum level) of E2 suppressed T cell activities, while lower dose E2 (postmenopausal serum level) activated T cell activity. The investigators have investigated the combination of anti-PD1 antibody and GnRH agonist plus exemestane (an aromatase inhibitor which will block the production of E2 from adipose tissue) in ER positive premenopausal breast cancer patient refractory to prior endocrine therapy in metastatic setting. The response rate was 38.4%, and median progression-free survival (PFS) was 10.2 months. This outstanding result were presented in AACR 2021 oral session (Cancer Res 2021 81:13_Supplement, CT028). On the other hand, progesterone is also well known for its anti-inflammation and immune tolerance activity. This possibly makes estrogen reduction treatments, such as gonadotropin-releasing hormone agonist (GnRH agonist), an important partner in augmenting neoadjuvant therapy for patients with premenopausal breast cancer.

For triple negative breast cancer (TNBC), endocrine therapy has no anti-tumor effect. On the other hand, the use of GnRH agonist has been tested for the protection of ovary function of young female while receiving adjuvant chemotherapy. Surprisingly, the concomitant use of goserelin and adjuvant chemotherapy improved disease-free survival (HR 0.47, P=0.04) and overall survival (HR 0.45, P=0.05) versus chemotherapy alone in ER negative premenopausal early BC patients in POEMS study, which was initially aimed to improve the success pregnant rate (N Engl J Med 2015 372;923). Endocrine therapy is theoretically antagonist to chemotherapy therapy when concomitantly use. In another report analyzed the outcome of both pre- and postmenopausal women who entered two randomized trials (Gruppo Oncologico Nord-Ovest-Mammella Intergruppo studies) on adjuvant chemotherapy and received either concomitant or sequential hormonal therapy. The result showed a decreasing trend (P = 0.015) in hazard ratio of death with increasing age was observed, indicating that concomitant therapy is more effective than sequential therapy in young patients (Annals of Oncology 2008;19(2):299-307). These results support the hypothesis that, E2 suppression/ER inhibition therapy may modulate immune microenvironment, thereby enhancing the chemotherapy induced immunogenic death effect.

The investigators hypothesized that, estrogen level reduction by ovarian function suppression can modulate immune microenvironment, thereby augmenting adjuvant chemotherapy efficacy, regardless of the estrogen receptor (ER) status of cancer cell. Therefore, the investigators plan to test this hypothesis in real clinical model, with standard clinical recommended treatment doses.

The study is designed to evaluate whether the GnRH agonist can provide the therapeutic benefit for premenopausal TNBC patients via modulating immune microenvironment. Premenopausal TNBC patients will receive GnRH agonist and neoadjuvant chemotherapy, and the efficacy and immune microenvironment change of co-administration arm will be measured and compared with chemotherapy alone control arm.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to fulfill all of the following criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Female patients aged ≥ 18 years at screening; Must be premenopausal according to serum E2, FSH level.
3. Histological confirmed TNBC, as defined by the most recent ASCO/CAP guidelines. Hormone receptor-low/HER2 negative as defined by ER 1% to <10% and/or PR 1% to <10% on IHC staining; neither hormone receptor may be ≥ 10%; and HER2-negative (IHC 0+/1+, or IHC 2+ plus FISH negative) is allowed.
4. Have previously untreated locally advanced non-metastatic (M0) TNBC and hormone receptor-low/HER2-negative defined as the following combined primary tumor (T) and regional lymph node (N) staging per current AJCC staging criteria for breast cancer staging criteria as assessed by the investigator based on radiological and/or clinical assessment: T1c, N0-N2; or T2, N0-N2; or T3, N0-N2; or T4a-d, N0-N2.
5. Agree to receive core needle biopsy for translational research.
6. ECOG 0-1.
7. Patients must have adequate organ and marrow reserve measured within 14 days prior to randomization as defined below:

   * Hemoglobin ≥ 9.0 g/dL;
   * Absolute neutrophil count ≥ 1,500 /μL;
   * Platelets ≥ 100,000/μL;
   * Total bilirubin ≤1.5 x upper normal limit;
   * AST(SGOT)/ALT(SGPT) ≤ 2.5 x upper normal limit;
   * Serum creatinine ≤ 1.5mg/dL or creatinine clearance ≧50ml/min;
   * aPTT < 1.5 x upper normal limit (unless on therapeutic anti-coagulation);
8. Plan to receive breast cancer surgery.
9. Must have a negative pregnancy test obtained within 3 days before starting therapy. Patients must not be breastfeeding.
10. Patients must use effective contraception prior to study entry and for the duration of study participation, and for 6 months after the completion of therapy.
11. Patients (or a surrogate) must be able to comply with study procedures and to give signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the clinical study protocol (CSP). The patients (or a surrogate) must be able to provide of signed and dated written ICF prior to any mandatory study specific procedures, sampling, and analyses.

Exclusion criteria Patients fulfilling any of the following criteria are not eligible for inclusion in this study. No additional exclusions may be applied by the Investigator, in order to ensure that the study population will be representative of all eligible patients.

1. Patients have received any prior therapy (including surgery, radiotherapy, chemotherapy, immunotherapy, or hormone therapy) for breast cancer.
2. Evidence of systemic metastasis.
3. Pregnancy or lactation.
4. Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
5. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs, with exception of hydroxychloroquine (Plaquenil®)) in subjects planning for pembrolizumab use.
6. Has a diagnosis of immunodeficiency or is receiving high dose of systemic steroid therapy. Patients with minor medical disease condition (i.e. mild asthma) requiring prednisolone equal to or less than 20 mg/day or the equivalent may be allowed.
7. Has an active systemic bacterial, viral or fungal infection requiring systemic therapy.
8. Psychiatric illness or social situation that would preclude study compliance.
9. Serious non-healing wound, ulcer, or bone fracture. Except for breast cancer related non-healing wound or ulcer.
10. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrolment.
11. History of allergic reaction to compounds of similar chemical composition to the study drugs.
12. Any of the following conditions or treatments that may impact the safety of the patient:

    * History of, or current, significant cardiac disease including cardiac failure (NYHA functional class II-IV), myocardial infarction (within 6 months), unstable angina (within 6 months), transient ischemic attack (within 6 months), stroke, cardiac arrhythmias requiring treatment or uncontrolled arterial hypertension
    * Concomitant clinically significant cardiac arrhythmias, e.g., sustained ventricular tachycardia, and clinically significant second- or third-degree AV block without a pacemaker on screening electrocardiogram (ECG)
    * History of or active severe respiratory disease, including Chronic Obstructive Pulmonary Disease, interstitial lung disease or pulmonary fibrosis
    * Severe hepatic impairment (Child-Pugh class C)
    * Any medically unstable condition as determined by the Investigator
13. Patients unable or unwilling to undergo serial breast tumor biopsy.
14. History of hypersensitivity to any of the study drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | During surgery
  No invasive residual in breast or nodes; non-invasive breast residuals allowed

SECONDARY OUTCOMES:
Event free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  To compare the event-free survival (EFS) assessed by investigator in ITT population after neoadjuvant chemotherapy with/without ovary suppression
Quality of life from patient-report outcome | At Screening phase, at Treatment 1 cycle 4 day 1 ( each cycle is 14 days or 21 days) , at Treatment 2 cycle 4 day 1 (each cycle is 14 days or 21 days), through study completion, an average of 5 years
  Quality of life will be assessed by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 , the minimum values is : 30 , the maximum values is : 126, the higher scores mean a worse outcome
Estradiol | At Screening phase, at Treatment 1 cycle 1 day 1, at Treatment 1 cycle 3 day 1, at Treatment 2 cycle 1 day 1, at Treatment 2 cycle 3 day 1, during surgery, through study completion, an average of 5 years
  Estradiol (E2) pg/mL
Follicle stimulating hormone | At Screening phase, at Treatment 1 cycle 1 day 1, at Treatment 1 cycle 3 day 1, at Treatment 2 cycle 1 day 1, at Treatment 2 cycle 3 day 1, during surgery, through study completion, an average of 5 years
  Follicle stimulating hormone (FSH) mIU/mL
Luteinizing hormone | At Screening phase, at Treatment 1 cycle 1 day 1, at Treatment 1 cycle 3 day 1, at Treatment 2 cycle 1 day 1, at Treatment 2 cycle 3 day 1, during surgery, through study completion, an average of 5 years
  Luteinizing hormone (LH) mIU/mL
Tumor microenvironment changes after neoadjuvant chemotherapy with/without ovarian suppression | At Screening phase, at Treatment 1 cycle 1 day 1 ( each cycle is 14 days or 21 days), at Treatment 2 cycle 1 day 1 ( each cycle is 14 days or 21 days), through study completion, an average of 5 years
  To evaluate the tumor-infiltrating lymphocytes (TIL)
Pathological complete response by tumor infiltrating lymphocyte | During surgery
  To evaluate the rate of pCR (ypT0/Tis ypN0) as assessed by the local pathologist at the time of definitive surgery in individuals with TIL(+) or TIL(-) tumors.
Residual cancer burden | During surgery
  To evaluate Residual Cancer Burden (RCB) as assessed by the local pathologist at the time of definitive surgery
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 32 weeks
  To determine the safety and tolerability of ovarian function suppression in combination with neoadjuvant chemotherapy in locally advanced TNBC subjects
Breast cancer quality of life from patient-report outcome | At Screening phase, at Treatment 1 cycle 4 day 1 ( each cycle is 14 days or 21 days) , at Treatment 2 cycle 4 day 1 ( each cycle is 14 days or 21 days), through study completion, an average of 5 years
  Breast cancer quality of life will be assessed by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire BR23 , the minimum values is : 22 , the maximum values is : 92, the higher scores mean a worse outcome
Event free survival by tumor infiltrating lymphocyte | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  To evaluate the event free survival by investigator in individuals with TIL(+) or TIL(-) tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin CH, Yap YS, Lee KH, Im SA, Naito Y, Yeo W, Ueno T, Kwong A, Li H, Huang SM, Leung R, Han W, Tan B, Hu FC, Huang CS, Cheng AL, Lu YS; Asian Breast Cancer Cooperative Group. Contrasting Epidemiology and Clinicopathology of Female Breast Cancer in Asians vs the US Population. J Natl Cancer Inst. 2019 Dec 1;111(12):1298-1306. doi: 10.1093/jnci/djz090. PMID 31093668
- [Background] Fan L, Strasser-Weippl K, Li JJ, St Louis J, Finkelstein DM, Yu KD, Chen WQ, Shao ZM, Goss PE. Breast cancer in China. Lancet Oncol. 2014 Jun;15(7):e279-89. doi: 10.1016/S1470-2045(13)70567-9. PMID 24872111
- [Background] Bauer KR, Brown M, Cress RD, Parise CA, Caggiano V. Descriptive analysis of estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, and HER2-negative invasive breast cancer, the so-called triple-negative phenotype: a population-based study from the California cancer Registry. Cancer. 2007 May 1;109(9):1721-8. doi: 10.1002/cncr.22618. PMID 17387718
- [Background] Dent R, Trudeau M, Pritchard KI, Hanna WM, Kahn HK, Sawka CA, Lickley LA, Rawlinson E, Sun P, Narod SA. Triple-negative breast cancer: clinical features and patterns of recurrence. Clin Cancer Res. 2007 Aug 1;13(15 Pt 1):4429-34. doi: 10.1158/1078-0432.CCR-06-3045. PMID 17671126
- [Background] Park YH, Senkus-Konefka E, Im SA, Pentheroudakis G, Saji S, Gupta S, Iwata H, Mastura MY, Dent R, Lu YS, Yin Y, Smruti BK, Toyama T, Malwinder S, Lee SC, Tseng LM, Kim JH, Kim TY, Suh KJ, Cardoso F, Yoshino T, Douillard JY. Pan-Asian adapted ESMO Clinical Practice Guidelines for the management of patients with early breast cancer: a KSMO-ESMO initiative endorsed by CSCO, ISMPO, JSMO, MOS, SSO and TOS. Ann Oncol. 2020 Apr;31(4):451-469. doi: 10.1016/j.annonc.2020.01.008. Epub 2020 Jan 16. PMID 32081575
- [Background] Liedtke C, Mazouni C, Hess KR, Andre F, Tordai A, Mejia JA, Symmans WF, Gonzalez-Angulo AM, Hennessy B, Green M, Cristofanilli M, Hortobagyi GN, Pusztai L. Response to neoadjuvant therapy and long-term survival in patients with triple-negative breast cancer. J Clin Oncol. 2008 Mar 10;26(8):1275-81. doi: 10.1200/JCO.2007.14.4147. Epub 2008 Feb 4. PMID 18250347
- [Background] Carey LA, Dees EC, Sawyer L, Gatti L, Moore DT, Collichio F, Ollila DW, Sartor CI, Graham ML, Perou CM. The triple negative paradox: primary tumor chemosensitivity of breast cancer subtypes. Clin Cancer Res. 2007 Apr 15;13(8):2329-34. doi: 10.1158/1078-0432.CCR-06-1109. PMID 17438091
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] von Minckwitz G, Untch M, Nuesch E, Loibl S, Kaufmann M, Kummel S, Fasching PA, Eiermann W, Blohmer JU, Costa SD, Mehta K, Hilfrich J, Jackisch C, Gerber B, du Bois A, Huober J, Hanusch C, Konecny G, Fett W, Stickeler E, Harbeck N, Muller V, Juni P. Impact of treatment characteristics on response of different breast cancer phenotypes: pooled analysis of the German neo-adjuvant chemotherapy trials. Breast Cancer Res Treat. 2011 Jan;125(1):145-56. doi: 10.1007/s10549-010-1228-x. Epub 2010 Nov 3. PMID 21042932
- [Background] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Background] Schmid P, Cortes J, Dent R, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Untch M, Fasching PA, Cardoso F, Andersen J, Patt D, Danso M, Ferreira M, Mouret-Reynier MA, Im SA, Ahn JH, Gion M, Baron-Hay S, Boileau JF, Ding Y, Tryfonidis K, Aktan G, Karantza V, O'Shaughnessy J; KEYNOTE-522 Investigators. Event-free Survival with Pembrolizumab in Early Triple-Negative Breast Cancer. N Engl J Med. 2022 Feb 10;386(6):556-567. doi: 10.1056/NEJMoa2112651. PMID 35139274
- [Background] Finn OJ. Cancer immunology. N Engl J Med. 2008 Jun 19;358(25):2704-15. doi: 10.1056/NEJMra072739. No abstract available. PMID 18565863
- [Background] Yarchoan M, Johnson BA 3rd, Lutz ER, Laheru DA, Jaffee EM. Targeting neoantigens to augment antitumour immunity. Nat Rev Cancer. 2017 Apr;17(4):209-222. doi: 10.1038/nrc.2016.154. Epub 2017 Feb 24. PMID 28233802
- [Background] Smith CC, Selitsky SR, Chai S, Armistead PM, Vincent BG, Serody JS. Alternative tumour-specific antigens. Nat Rev Cancer. 2019 Aug;19(8):465-478. doi: 10.1038/s41568-019-0162-4. Epub 2019 Jul 5. PMID 31278396
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Versluis JM, Long GV, Blank CU. Learning from clinical trials of neoadjuvant checkpoint blockade. Nat Med. 2020 Apr;26(4):475-484. doi: 10.1038/s41591-020-0829-0. Epub 2020 Apr 9. PMID 32273608
- [Background] Liu J, Blake SJ, Yong MC, Harjunpaa H, Ngiow SF, Takeda K, Young A, O'Donnell JS, Allen S, Smyth MJ, Teng MW. Improved Efficacy of Neoadjuvant Compared to Adjuvant Immunotherapy to Eradicate Metastatic Disease. Cancer Discov. 2016 Dec;6(12):1382-1399. doi: 10.1158/2159-8290.CD-16-0577. Epub 2016 Sep 23. PMID 27663893
- [Background] Blank CU, Rozeman EA, Fanchi LF, Sikorska K, van de Wiel B, Kvistborg P, Krijgsman O, van den Braber M, Philips D, Broeks A, van Thienen JV, Mallo HA, Adriaansz S, Ter Meulen S, Pronk LM, Grijpink-Ongering LG, Bruining A, Gittelman RM, Warren S, van Tinteren H, Peeper DS, Haanen JBAG, van Akkooi ACJ, Schumacher TN. Neoadjuvant versus adjuvant ipilimumab plus nivolumab in macroscopic stage III melanoma. Nat Med. 2018 Nov;24(11):1655-1661. doi: 10.1038/s41591-018-0198-0. Epub 2018 Oct 8. PMID 30297911
- [Background] Hamilton DH, Griner LM, Keller JM, Hu X, Southall N, Marugan J, David JM, Ferrer M, Palena C. Targeting Estrogen Receptor Signaling with Fulvestrant Enhances Immune and Chemotherapy-Mediated Cytotoxicity of Human Lung Cancer. Clin Cancer Res. 2016 Dec 15;22(24):6204-6216. doi: 10.1158/1078-0432.CCR-15-3059. Epub 2016 Jun 7. PMID 27267852
- [Background] Svoronos N, Perales-Puchalt A, Allegrezza MJ, Rutkowski MR, Payne KK, Tesone AJ, Nguyen JM, Curiel TJ, Cadungog MG, Singhal S, Eruslanov EB, Zhang P, Tchou J, Zhang R, Conejo-Garcia JR. Tumor Cell-Independent Estrogen Signaling Drives Disease Progression through Mobilization of Myeloid-Derived Suppressor Cells. Cancer Discov. 2017 Jan;7(1):72-85. doi: 10.1158/2159-8290.CD-16-0502. Epub 2016 Sep 30. PMID 27694385
- [Background] Moore HC, Unger JM, Phillips KA, Boyle F, Hitre E, Porter D, Francis PA, Goldstein LJ, Gomez HL, Vallejos CS, Partridge AH, Dakhil SR, Garcia AA, Gralow J, Lombard JM, Forbes JF, Martino S, Barlow WE, Fabian CJ, Minasian L, Meyskens FL Jr, Gelber RD, Hortobagyi GN, Albain KS; POEMS/S0230 Investigators. Goserelin for ovarian protection during breast-cancer adjuvant chemotherapy. N Engl J Med. 2015 Mar 5;372(10):923-32. doi: 10.1056/NEJMoa1413204. PMID 25738668
- [Background] Del Mastro L, Dozin B, Aitini E, Catzeddu T, Baldini E, Contu A, Durando A, Danese S, Cavazzini G, Canavese G, Bruzzi P, Pronzato P, Venturini M; GONO-MIG Group. Timing of adjuvant chemotherapy and tamoxifen in women with breast cancer: findings from two consecutive trials of Gruppo Oncologico Nord-Ovest-Mammella Intergruppo (GONO-MIG) Group. Ann Oncol. 2008 Feb;19(2):299-307. doi: 10.1093/annonc/mdm475. Epub 2007 Oct 17. PMID 17947224
- [Background] West CP, Baird DT. Suppression of ovarian activity by Zoladex depot (ICI 118630), a long-acting luteinizing hormone releasing hormone agonist analogue. Clin Endocrinol (Oxf). 1987 Feb;26(2):213-20. doi: 10.1111/j.1365-2265.1987.tb00779.x. PMID 2959405
- [Background] Francis PA, Pagani O, Fleming GF, Walley BA, Colleoni M, Lang I, Gomez HL, Tondini C, Ciruelos E, Burstein HJ, Bonnefoi HR, Bellet M, Martino S, Geyer CE Jr, Goetz MP, Stearns V, Pinotti G, Puglisi F, Spazzapan S, Climent MA, Pavesi L, Ruhstaller T, Davidson NE, Coleman R, Debled M, Buchholz S, Ingle JN, Winer EP, Maibach R, Rabaglio-Poretti M, Ruepp B, Di Leo A, Coates AS, Gelber RD, Goldhirsch A, Regan MM; SOFT and TEXT Investigators and the International Breast Cancer Study Group. Tailoring Adjuvant Endocrine Therapy for Premenopausal Breast Cancer. N Engl J Med. 2018 Jul 12;379(2):122-137. doi: 10.1056/NEJMoa1803164. Epub 2018 Jun 4. PMID 29863451
- [Background] Garcia-Giralt E, Beuzeboc P, Dieras V, Dorval T, Jouve M, Livartowski A, Palangie T, Scholl S, Pouillart P. Phase II trial of decapeptyl (D-TRP-6), a potent luteinizing hormone-releasing hormone analogue in untreated advanced breast cancer. Am J Clin Oncol. 1996 Oct;19(5):455-8. doi: 10.1097/00000421-199610000-00006. PMID 8823473
- [Background] Pagani O, Regan MM, Walley BA, Fleming GF, Colleoni M, Lang I, Gomez HL, Tondini C, Burstein HJ, Perez EA, Ciruelos E, Stearns V, Bonnefoi HR, Martino S, Geyer CE Jr, Pinotti G, Puglisi F, Crivellari D, Ruhstaller T, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Bernhard J, Luo W, Ribi K, Viale G, Coates AS, Gelber RD, Goldhirsch A, Francis PA; TEXT and SOFT Investigators; International Breast Cancer Study Group. Adjuvant exemestane with ovarian suppression in premenopausal breast cancer. N Engl J Med. 2014 Jul 10;371(2):107-18. doi: 10.1056/NEJMoa1404037. Epub 2014 Jun 1. PMID 24881463
- [Background] Nanda R, Liu MC, Yau C, Shatsky R, Pusztai L, Wallace A, Chien AJ, Forero-Torres A, Ellis E, Han H, Clark A, Albain K, Boughey JC, Jaskowiak NT, Elias A, Isaacs C, Kemmer K, Helsten T, Majure M, Stringer-Reasor E, Parker C, Lee MC, Haddad T, Cohen RN, Asare S, Wilson A, Hirst GL, Singhrao R, Steeg K, Asare A, Matthews JB, Berry S, Sanil A, Schwab R, Symmans WF, van 't Veer L, Yee D, DeMichele A, Hylton NM, Melisko M, Perlmutter J, Rugo HS, Berry DA, Esserman LJ. Effect of Pembrolizumab Plus Neoadjuvant Chemotherapy on Pathologic Complete Response in Women With Early-Stage Breast Cancer: An Analysis of the Ongoing Phase 2 Adaptively Randomized I-SPY2 Trial. JAMA Oncol. 2020 May 1;6(5):676-684. doi: 10.1001/jamaoncol.2019.6650. PMID 32053137